CLINICAL TRIAL: NCT04991415
Title: Manual Therapy for the Treatment of Shoulder Pain for Overuse Syndrome Wheelchair Dependent Persons
Acronym: MTX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Coker, Research Scientist I, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Manual Therapy
Record Dates: First submitted 2016-09-20; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Spinal Cord Injuries; Pain; Musculoskeletal Manipulations
MeSH Terms: conditions — Spinal Cord Injuries; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): 30 minutes of manual therapy three times a week for two weeks (six total sessions).
  Interventions: Other: Manual Therapy
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Manual Therapy
  Arms: Treatment

SUMMARY:
Shoulder pain is a common, debilitating problem for persons with Spinal cord injuries (SCI). Shoulder pain affects approximately 40-50% of the total population of persons with paraplegia (those with SCI with full use of their upper extremities and no or limited use of their lower extremities). Among the etiologies of shoulder pain in persons with paraplegia, overuse syndrome is the most common. Shoulder overuse syndrome in a person with paraplegia is the result of high activity demands and high mechanical load on the upper extremity during activities such as wheelchair propulsion, transferring with the arms, and performing activities of daily living from a wheelchair height, resulting in increased overhead activity. The pain as a result of overuse syndrome can limit the patient's participation in occupational and physical therapy as well as limit performance of activities of daily living and participation in usual life activities. An alternative treatment for shoulder pain with evidence to support efficacy in the able bodied population is Manual Therapy (MT). Unfortunately, there have been no prior research studies published examining the therapeutic efficacy of MT for overuse injuries of the shoulder in patients with paraplegia. This study will determine if MT, is efficacious to reduce pain in this population. A total of 20 patients with paraplegia identified in the outpatient clinic at Craig Hospital with overuse syndrome of the shoulder will be enrolled in the study.

DETAILED DESCRIPTION:
Shoulder pain is a common, debilitating problem for persons with Spinal cord injuries (SCI). Shoulder pain affects approximately 40-50% of the total population of persons with paraplegia (those with SCI with full use of their upper extremities and no or limited use of their lower extremities). Among the etiologies of shoulder pain in persons with paraplegia, overuse syndrome is the most common. Shoulder overuse syndrome in a person with paraplegia is the result of high activity demands and high mechanical load on the upper extremity during activities such as wheelchair propulsion, transferring with the arms, and performing activities of daily living from a wheelchair height, resulting in increased overhead activity. The pain as a result of overuse syndrome can limit the patient's participation in occupational and physical therapy as well as limit performance of activities of daily living and participation in usual life activities.

In the able bodied population, the most common recommendation for overuse syndrome is resting the affected joint. In persons with paraplegia and wheelchair dependence, this recommendation is unrealistic and would lead to non-use of the person's primary means of mobility (the wheelchair). Often, patients require pharmacologic intervention to help alleviate the pain in order to participate in therapy sessions and activities of daily living. Current treatment options for overuse syndrome include oral medication including narcotic pain medication and anti-inflammatory medication, modalities, injections, and surgery. Despite these treatment options, pain from overuse syndrome remains a prevalent problem with no treatment option proven superior and no gold standard of treatment identified. An alternative treatment for shoulder pain with evidence to support efficacy in the able bodied population is Manual Therapy (MT). Unfortunately, there have been no prior research studies published examining the therapeutic efficacy of MT for overuse injuries of the shoulder in patients with paraplegia. This study will determine if MT, is efficacious to reduce pain in this population. A total of 20 patients with paraplegia identified in the outpatient clinic at Craig Hospital with overuse syndrome of the shoulder will be enrolled in the study. Ten of the participants will be randomized to the control group and receive no MT and ten participants will be randomized to the treatment group and receive MT for three days per week x 2weeks. The treatment will be provided by a Doctor of Osteopathic Medicine (D.O.), physical, or occupational therapists trained to perform MT. During this study, the subject's pain and function will be measured by a 10 point questionnaire, the Numeric Pain Rating Scale (NPRS) and the Wheelchair Users Shoulder Pain Index (WUSPI). The NPRS and WUSPI are included in Appendix 1 and 2. The NPRS has been validated as a ratio scale for pain. The WUSPI has been validated as a scale for assessment of baseline shoulder dysfunction and for periodic measurement in longitudinal studies of musculoskeletal complications in wheelchair users. Data gathered from these outcome measures will be accumulated and statistically analyzed to examine the potential benefit of MT in the target population. This investigation will be one of the first to examine the relationship between MT and reduction in shoulder pain for treatment of overuse syndrome in persons with paraplegia. It will also examine if decreased pain secondary to MT will result in a decrease in pain during functional activity in these individuals. The results of this pilot study may result in publication in peer reviewed journals, presentations at national symposiums and application for funding for Complementary Medicine grant by the National Institute of Health or other available grant for larger study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65,
* Spinal cord injury, non-ambulatory, wheelchair user,
* Pain in shoulder from overuse injury,
* Pain interference on the WUSPI of at least 6/10 on at least 2 of the transfer items and any one of the remaining items,
* English-speaking,
* Stable spine,
* Full weight-bearing status in bilateral upper extremities (i.e. no orthopedic precautions on UE weight-bearing activities)
* Greater than 3 months post initial spinal cord injury
* Diagnosis of overuse syndrome of the shoulder

Exclusion Criteria:

* Concomitant moderate to severe Traumatic Brain Injury
* Fractures in upper limbs.
* Concurrent diagnosis of Fibromyalgia.
* Cervical radiculopathy.
* Previous shoulder pathology
* Neuromuscular junction disorders (such as myasthenia gravis),
* Psychiatric disorder.
* Lack capacity to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Change in Wheelchair Users Shoulder Pain Index (WUSPI) | Two weeks
  WUSPI collected at baseline (before treatment) and two weeks (after treatment)

SECONDARY OUTCOMES:
Change in Numerical Pain Rating Scale (NPRS) | Two weeks
  NPRS collected at baseline (before treatment) and two weeks (after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Berliner, DO, Principal Investigator — Physician, Director of Outpatient Medicine
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided